### **Participant Informed Consent for Clinical Research**

**Study title for participants:** A Study on Radiation Therapy Guided by the Reflectance Confocal Microscopy (RCM)/Optical Coherence Tomography (OCT) Device in People with Basal Cell Carcinoma

Official study title for internet search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>: A Phase II Trial of Reflectance Confocal Microscopy and Optical Coherence Tomography Guided Radiation Therapy: CLARITY

**Lead Researcher:** Christopher Barker, MD (212-639-8168)

If you are the legally authorized representative (LAR) of the person who is being asked to participate in this research study, you may give consent on his or her behalf. The word "you" in this document refers to the study participant.

## **Overview and Key Information**

### Why is this study being done?

We are asking you to take part in a clinical research study. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

You are being asked to take part in this research study because you have basal cell carcinoma (BCC), and you are planning to have radiation therapy (RT) to treat your skin cancer.

The most effective treatment for BCC is surgery, but this might not be an option for or the preference of all patients. The most effective non-surgical option is RT. A challenge with RT is being able to see all of the cancer cells that need to be treated. Sometimes doctors have difficulty with being able to see which cells are cancerous and which ones are healthy. In addition, it can be hard to see if any cancer remains after RT. If cancer cells remain after RT, surgery may be needed to remove those cells.

Reflectance confocal microscopy (RCM) and optical coherence tomography (OCT) are two imaging tools routinely used to identify the presence of skin cancer. RCM uses a laser to see which cells are healthy and which cells are cancerous and identify the outer edges of the tumor (the margin). OCT uses near-infrared light (invisible and deeply penetrating light) to see how deep cancer cells go.

Researchers think that combining these two imaging tools into one device (the RCM/OCT device) and using that device to guide RT could help with the treatment of BCC. We are doing this study to find out if RT guided by the RCM/OCT device is an effective treatment for BCC.

The US Food and Drug Administration (FDA) has approved RT for the treatment of BCC and has approved the RCM and OCT as separate devices to help diagnose skin cancer. The FDA has not approved the new combined RCM/OCT device for use with RT, or any other purposes, but researchers are permitted to test it in studies like this one. The use of the RCM/OCT device in this study is considered investigational.

## Taking part in this study is your choice.



You can choose to take part or not to take part in this study, and you can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document presents important information to help you make your choice. Please take time to read it carefully. Talk with your doctor, family, or friends about the risks and benefits of taking part in this study. It's important that you have as much information as you need, and that all your questions are answered.

### What is the usual approach to treating BCC?

People with BCC can have a variety of treatments for their skin cancer. Surgery is the most common treatment, but other non-surgical treatments can be considered, with RT being considered the most effective. After non-surgical treatments (like RT), a repeat biopsy is routinely done to see if any cancer cells remain. If there are remaining cancer cells, the usual approach is to perform surgery to remove the cells.

## What are my other choices if I decide not to take part in this study?

- You may choose to have the usual approach described above
- You may choose to take part in a different research study, if one is available
- You may choose not to be treated for cancer

## What will happen if I decide to take part in this study?

If you decide to participate in this study, we will look at your tumor using the RCM/OCT device, and then you will have the standard RT for your BCC. The RCM/OCT device is a handheld device that the study doctor will hold over your area of BCC.

Six weeks after your RT, you will come back to the clinic to have your tumor looked at using the RCM/OCT device again. You will also have a routine biopsy to see if any cancer cells remain. If cancer cells are found in your biopsy sample, you may have surgery as part of your routine care to remove the remaining cells. Your study doctor will discuss treatment options with you.

Starting 20 weeks after RT, we will review your medical records, and we may call you, email you, or mail you a letter every 6 months for up to 3 years to check on your health and BCC.

## What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important to think carefully about these as you make your decision.

#### Ricks

We want to make sure that you know about a few key risks right now. We will also give you more information in the *What risks can I expect from taking part in this study?* section of this consent form.

If you choose to take part in this study, there is a risk that the study approach may not be any better than the usual approach of having RT without use of an imaging tool.

There is also a risk that you could have side effects from the study approach. These side effects may be worse, and they may be different than you would have with the usual approach for your cancer.

There are no known risks of using the RCM/OCT device.



Some of the most common side effects of RT that the study doctors know about are:

- Swelling, redness, itchiness, thinning, hardening, darkening, or lightening of the treated area on the skin
- Pain
- Hair loss
- Spider veins (small, twisted blood vessels that are visible through the skin)

There may be some risks that the study doctors do not yet know about.

#### **Benefits**

RT with and without use of RCM and OCT has been shown to treat and cure your type of cancer. It is not possible to know now if RT guided by the new RCM/OCT device will be effective. Your cancer may get better, or it may stay the same or get worse. What we learn from this study may help other people in the future.

### If I decide to take part in this study, can I stop later?

Yes, you can decide to stop participating in the study at any time.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

If you decide to stop, let the study doctor know as soon as possible. It's important that you stop safely.

If you stop, you can decide whether to let the study doctor or a member of the study team continue to contact you to ask questions about your health. We will not be able to withdraw information about you that has been used or shared with others before you informed us of your decision to stop.

## Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes, and the study is no longer in your best interest
- New information becomes available, and the study is no longer in your best interest
- You do not follow the study rules
- For women who are able to have children: You become pregnant while you are in the study
- The study is stopped by the National Cancer Institute (NCI), Institutional Review Board (IRB), US Food and Drug Administration (FDA), or the study sponsor, Memorial Sloan Kettering Cancer Center (MSK). The study sponsor is the organization that oversees the study.

It is important that you understand the information in this informed consent document before you make a decision about participating in this clinical trial. Please read, or have someone read to you, the rest of this document. If there is anything that you don't understand, ask the study doctor or nurse for more information.

## What is the purpose of this study?

The purpose of this study is to find out if radiation therapy (RT) guided by the new reflectance confocal microscopy (RCM)/optical coherence tomography (OCT) device is an effective treatment for basal cell



Memorial Sloan Kettering Cancer Center IRB Number: 20-553 A(7) Approval date: 18-Mar-2024

carcinoma (BCC). We will also look at the side effects from RT guided by the RCM/OCT device. In addition, we will determine your quality of life before and after their treatment by having you fill out questionnaires.

Researchers think that combining the standard RCM and OCT imaging tools into one device (the RCM/OCT device) and using that device to guide RT could help with the treatment of BCC. RCM allows doctors to see which cells are healthy and which cells are cancerous and identify the outer edges of the tumor (the margin). OCT can show how deep cancer cells go. By combining RCM with OCT in one device, doctors may be able to get a fuller view of the tumor. Using the device to guide RT may help the RT be more precise in killing cancer cells and sparing healthy cells. Use of the RCM/OCT device may also help prevent the need for additional treatments, such as surgery. In addition, because the device may help the RT be more precise, less radiation may be used during the RT, and this decreased amount of radiation may cause side effects to be less frequent and less severe.

The US Food and Drug Administration (FDA) has approved RT for the treatment of BCC and has approved the RCM and OCT as separate devices to help diagnose skin cancer. The FDA has not approved the new combined RCM/OCT device for use with RT, or any other purposes, but researchers are permitted to test it in studies like this one. The use of the RCM/OCT device in this study is considered investigational.

The RCM/OCT device will be provided by Physical Sciences Inc.

About 38 people will take part in this study at Memorial Sloan Kettering Cancer Center (MSK).

## What are the study groups?

All participants will receive RT and have their tumor looked at using the RCM/OCT device.

## What extra tests and procedures will I have if I take part in this study?

#### Before you begin the main part of the study:

The study doctor will review your medical records and the results of your exams, tests, and procedures to see if it is safe for you to take part in the study. This first part of the study is called screening. Most of the screening exams, tests, and procedures are part of the usual care that you would have if you were not in a study.

The tests and procedures that will be done only for research purposes, or that may be done more often because you are participating in this study, are listed below.

You will complete questionnaires about how your skin cancer is affecting your quality of life.
 These questionnaires will be on paper, and they will take about 5-10 minutes to complete.

#### **During the study:**

At your Day 0 visit, we will take pictures of your BCC using a digital camera, and we will look at your tumor using the RCM/OCT device. The RCM/OCT device is a handheld device that the study doctor will hold over your area of BCC. We will use a pen to mark the borders of your BCC.

After we use the RCM/OCT device on you, you will start your RT. You will come to the clinic for RT over a period of up to 4 weeks. Your study doctor will let you know how many RT sessions you need to have.



Six weeks after the RT, you will come back to the clinic to have your tumor looked at again using the RCM/OCT device. You will also have a routine biopsy to see if any cancer cells remain. If cancer cells are found in your biopsy sample, you may have surgery as part of your routine care to remove the remaining cells. Your study doctor will discuss treatment options with you.

#### Exams, Tests, and/or Procedures

You will have exams, tests, and/or procedures during the main study. The procedures that will be done only for research purposes, or that may be done more often because you are participating in this study, are listed below.

You will complete quality-of-life questionnaires at every visit; 2, 6, and 12 weeks after you complete RT.

#### Follow-up:

Starting 20 weeks after you finish RT, we will review your medical records, and we may call you, email you, or mail you a letter every 6 months for up to 3 years to check on your health and BCC.

A Study Calendar that shows how often you will have these exams, tests, and procedures is provided at the end of this consent form. The calendar also includes exams, tests, and procedures that are part of your usual care.

#### Will I receive the results of my research tests?

You will not have any tests done for research purposes during this study. You will not receive the general results of this research study.

## What risks can I expect from taking part in this study?

If you choose to take part in this study, there is a risk that:

- You may lose time at work, school, or at home, and you may spend more time than usual in the hospital or doctor's office
- You may be asked sensitive or private questions that you do not usually discuss

The study intervention used in this study may affect how your skin looks or works. The study doctor will let you know if changes occur that may affect your health.

There is also a risk that you could have side effects from the study approach.

Important information about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, and some may never go away.
- Some side effects may make it difficult for you to have children.
- Some side effects may be mild. Others may be very serious, and may even result in death.

Important information about how you and the study doctor can make side effects less of a problem for you:

- If you notice or feel anything different, tell the study doctor. He or she can check to see if you are having a side effect.
- The study doctor may be able to treat some side effects.



The tables below show the most common and the most serious side effects that researchers know about. There may be other side effects that the doctors do not yet know about. If important new side effects are found during this study, the study doctor will discuss them with you.

There are no known risks of using the RCM/OCT device.

#### Possible side effects of radiation therapy:

#### Common, some may be serious

In 100 people receiving radiation therapy, more than 20 and as many as 100 may have:

- Skin changes, including swelling, redness, itchiness, thinning, hardening, darkening, or lightening of the treated area on the skin
- Spider veins (small, twisted blood vessels that are visible through the skin)
- Permanent hair loss in the area treated with radiation
- Pain

#### Rare, and serious

In 100 people receiving radiation therapy, 3 or fewer may have:

A new cancer develops at the treated site

**Reproductive risks**: You should not get pregnant, breastfeed, father a baby, or donate sperm while you are in this study. The radiation therapy used in this study could be very damaging to an unborn baby. Check with the study doctor about what types of birth control or pregnancy prevention to use while you are in this study. You must continue to use these methods for 1 year after completing the study treatment.

Let the study doctor know about any questions you may have about possible side effects. You can ask the study doctor questions about side effects at any time.

## What are my responsibilities in this study?

If you choose to take part in this study, you will need to:

- Keep your study appointments
- Tell the study doctor about:
  - All medications and any supplements you are taking
  - Any side effects from these medications or supplements
  - Any doctor visits or hospital stays outside of this study
  - Whether you have been or are currently in another research study
- Let the study doctor know if you skipped or chose not to answer any of the questions in the questionnaire/survey.

## Is there a conflict of interest for this study?

This study is sponsored by Memorial Sloan Kettering Cancer Centers with support provided by the National Institutes of Health (NIH) and Physical Sciences Inc. One of the investigators involved in this study has a financial interest which might be affected by the results of the study. This means that the investigator could gain or lose money, depending on the results of the study.



If you would like to know more about the steps MSK has taken to protect your best interests while you are in this study, please contact the MSK Patient Representative Department at 212-639-7202.

## What are the costs of taking part in this study?

You will not have to pay for the use of the RCM/OCT device.

You and/or your health plan/insurance company will have to pay for all the other costs of treating your cancer while you are in this study. These charges include the costs of RT, insurance co-pays and deductibles, as well as tests, procedures, or drugs that you get during the study to monitor your safety, and to prevent or manage any side effects.

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it does not pay for if you take part in this clinical trial. Also find out if you need approval from your health plan before you can take part in this study.

The study doctor or nurse can help you find the right person to talk to if you are not sure which costs will be billed to you or your insurance provider.

## Will I receive payment for taking part in this study?

You will not be paid for taking part in this study.

## What happens if I am injured or hurt because I took part in this study?

You will get medical treatment if you are injured as a result of taking part in this study.

If you think that you have been injured as a result of taking part in this research study, tell the study doctor or the person in charge of the study as soon as possible. The name and telephone number of the person in charge of this research are listed on the first page of this consent form.

We will offer you treatment for research injuries that happen as a result of your taking part in this study. You and/or your health plan will be charged for this treatment. Medical services will be offered at the usual charge. You will be responsible for any costs not covered by your health plan/insurance company.

If you think that your injury was a result of medical error, you keep all your legal rights to receive payment for treating the injury, even though you are in a study.

## Who will see my medical information?

Your privacy is very important to us, and the researchers will make every effort to protect it. Trained staff at Memorial Hospital may review your records, if necessary.

Access to your protected health information will be limited to those listed in the Research Authorization form, which is a part of the informed consent process.

Your information may be given out, if required by law. For example, some states require doctors to make a report to the state health board if they find that a participant in a research study has a contagious disease like tuberculosis. However, the researchers will do their best to make sure that any information about you that may be released will not identify you.



Memorial Sloan Kettering Cancer Center IRB Number: 20-553 A(7) Approval date: 18-Mar-2024

In the future, your information (data) may be de-identified, which means that your data will be assigned a unique code, and the list that links the code to your name will be stored separately from your data. Your de-identified information may be used for research that has not been described in this consent form, and they may be shared with another investigator for future research. You will not be asked if you agree to take part in future research studies.

If your information from this study is used in any reports or publications, your name and anything else that could identify you will not be used. It is possible that your de-identified information from this study will be shared with other researchers outside of MSK, and may be stored in public databases related to research. All requests for data sharing will be reviewed by the study sponsor, and if individual results are included in the data, they will not contain any identifiable information about you, such as your name, address, telephone number, or Social Security number. Your privacy is very important to us and we use many safety procedures to protect your privacy. However, we cannot guarantee that no one will ever be able to use your information to identify you.

The study doctors have a Certificate of Confidentiality from the National Institutes of Health for this study. This gives MSK an additional way to protect sensitive information that identifies you in your records if it is requested as part of a legal proceeding. However, MSK may still be required to share some of your medical information if required by law.

### Where can I get more information?

You may visit the NCI web site at <a href="http://cancer.gov/">http://cancer.gov/</a> for more information about research studies, or for general information about cancer. You may also call the NCI Cancer Information Service to get the same information at 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can talk to the study doctor about any questions or concerns that you may have about this study, or to report side effects or injuries. You may also contact the lead researcher listed on the first page of this consent.

For questions about your rights while you are participating in this study, call the MSK Institutional Review Board (IRB) at 212-639-7592. If you have concerns, complaints, or input on research, or if you would like more information about the informed consent process, please contact the MSK Patient Representative Department at 212-639-7202.



## Research Authorization for the Use and Disclosure of Protected Health Information (PHI)

A Study on Radiation Therapy Guided by the Reflectance Confocal Microscopy (RCM)/Optical Coherence Tomography (OCT) Device in People with Basal Cell Carcinoma

Federal law requires Memorial Sloan Kettering Cancer Center (MSK) to protect the privacy of information that identifies you and relates to your past, present, and future medical conditions (protected health information; PHI). We are committed to protecting the privacy of your information.

If you enroll in this research study, your protected health information will be used and shared with others, as explained below. MSK must obtain your permission before using or sharing your protected health information for research purposes. This form helps to make sure that you are informed of the ways in which your information will be used or shared in the future.

Carefully read the information below before you sign this form. By signing this form, you agree to the use and disclosure of your information for this research study.

# 1. What protected health information about me will be used or shared with others during this research?

- Your medical records
- Your research records, including new health information created from study-related tests, procedures, visits, and/or questionnaires
- Any health information or clinical data associated with your biospecimens, if the information or data could be reasonably used to identify you. This information or data will be shared only if you have agreed to it by signing this informed consent document.
- HIV-related information, including any information indicating that you have had an HIV-related test; or that you have HIV infection, HIV-related illness, or AIDS; or any information that could indicate that you may have been exposed to HIV. (New York State requires us to obtain your consent to use or share this information.)

## 2. Who will use or share my protected health information?

MSK will use and share your protected health information. People and offices that deal with research oversight, quality assurance, and/or billing will be able to use and share your protected health information, including:

- The study's Principal Investigator and Co-Principal Investigators: Christopher Barker, MD; Chih-Shan Chen, MD, PhD; and Anthony Rossi, MD
- Your research team at MSK, including the participating investigators, research staff, research nurses, fellows/residents, and clerical support staff
- Any healthcare personnel who provide services to you in connection with this study
- Members and staff of MSK's Institutional Review Board (IRB) and Privacy Board (PB)
- Staff of MSK's Clinical Research Administration, which oversees clinical studies, and Clinical Research Information Technology Group, which manages research databases
- Members of MSK's Data Safety Monitoring Board/Committee and the Quality Assurance Committee



IRB Number: 20-553 A(7) Approval date: 18-Mar-2024

## 3. With whom outside of MSK may my protected health information be shared?

Although all reasonable efforts will be made to maintain the confidentiality of your protected health information, it may be shared with and used by the following:

- The company and organization that provide the funding for the study, Physical Sciences Inc. and National Institutes of Health (NIH).
- MSK's research collaborators, business partners, subcontractors and agent(s), in the United States or in other countries, working to conduct the study, to monitor the study, or to analyze the study information for this study or for other research about the study device.
- Other research doctors and medical centers participating in this research.
- Federal and state agencies, and other domestic or foreign government bodies, if required by law and/or necessary for oversight purposes, including:
  - Office for Human Research Protections (OHRP) of the US Department of Health and Human Services (HHS)
  - US Food and Drug Administration (FDA) and other regulatory agencies responsible for oversight of research
  - National Cancer Institute (NCI)/National Institutes of Health (NIH)
- Other qualified researchers, approved by MSK, who may receive individual research results that do not identify you.

Some of the organizations that may receive your protected health information may not have to satisfy the privacy rules and requirements; they may share your information with others without your permission.

## 4. Why will my protected health information be used by or shared by MSK or others?

The main reasons for the use or sharing of your information include the following:

- To conduct the study, to monitor your health status, to measure the effects of the drug(s)/device(s)/procedure(s) being studied, and to determine the research results
- To ensure that the research meets legal and institutional requirements
- To develop new tests, procedures, and commercial products
- To enhance research databases, so that scientists can design better research studies to develop new therapies for patients and to gain a better understanding of disease
- To assist with MSK medical treatment, billing, or healthcare operations. For example, medical information produced by this research study will become part of your hospital medical record.

## 5. For how long will my protected health information be used or shared with others?

There is no set date at which your protected health information that is being used or shared for this research study will be destroyed or no longer used. The information used and created during the



Memorial Sloan Kettering Cancer Center IRB Number: 20-553 A(7)
Approval date: 18-Mar-2024

study may be analyzed for many years, and it is not possible to know when this analysis will be completed.

## 6. Statement of privacy rights:

- It is your right to refuse to sign this authorization form. If you do not sign this form, you will not be able to participate in this research study. However, if you do not sign, it will not affect your ongoing medical treatment or healthcare coverage.
- You have the right to withdraw your permission for MSK to use or share your protected health information. Please note that we will not be able to withdraw all the information about you that already has been used or shared with others to carry out research-related activities such as oversight, or information that is needed to ensure the quality of the study. To withdraw your permission, write to the study doctor listed on the first page of this consent form at: Memorial Sloan Kettering Cancer Center, 1275 York Avenue, New York, NY 10065. If you withdraw permission for us to use or share your protected health information, you will not be able to continue to participate in this research study.
- You have the right to request access to your protected health information that is being used or shared during this research and that is related to the research or to payment for the research. However, you may access this information only after the study is completed. You may have access to the parts of your medical record that are unrelated to this study at any time. To request this information, please contact the study doctor whose name and telephone number are listed on the first page of this consent form. You may also ask the study doctor to correct any study-related information about you that is wrong.

#### **Notice concerning HIV-related information**

Individuals/organizations are prohibited from sharing any HIV-related information about you without your approval, unless they are permitted to do so under federal or state law. You have a right to request the list of people who may receive or use your HIV-related information without your authorization.

If you experience discrimination because of the release or disclosure of your HIV-related information, you may contact the New York State Division of Human Rights at 888-392-3644 or the New York City Commission on Human Rights at 212-306-7500. These agencies are responsible for protecting your rights.



Memorial Sloan Kettering Cancer Center IRB Number: 20-553 A(7)
Approval date: 18-Mar-2024

## Participant Informed Consent/Research Authorization for Clinical Research Statement of professional obtaining consent

I have fully explained this clinical research study to the participant or to his/her Legally Authorized Representative (LAR). In my judgment, and in that of the participant or his/her LAR, sufficient information, including risks and benefits, was provided for the participant or his/her LAR to make an informed decision. The consent discussion will be documented in the participant's EMR.

Consenting professional must personally sign and date

| Consenting professiona | l's | | Date: |
|---|---|---|---|
| signature | | | |
| Consenting professiona (Print) | l's name | | |
| Participant's (or Legally Authorized Representative's [LAR's)]) statement I have read this form that describes the clinical research study. I have also talked it over to my satisfaction with the consenting professional. By signing below, I agree to the following: (1) to voluntarily participate in this clinical research study; (2) to authorize the use and disclosure of my/the participant's protected health information (data about myself/the participant); and (3) to state that I have received a signed and dated copy of this consent form. | | | |
| Participant/LAR must personally sign and date | | | |
| Participant/LAR | | Dat | æ: |
| signature | | | |
| Participant/LAR | | · | |
| name (Print) | | | |

| participant | | |
|---|---|---|
| Witness signature (if red | <u>quired)</u> | |
| ☐ Witness for non-English speaking participant: I declare that I am fluent in both English and in the participant's (or LAR's) language, and I confirm that the consent discussion was appropriately interpreted for the participant (or LAR). | | |
| Other: I confirm that the consent discussion occurred, and that the participant agreed to participate in this study by signing this form, making his/her mark, or verbally agreeing. | | |
| Name of witness: | | |
| Signature of witness: | | Date: |
| (The name of the witness must | t be documented in the EMR.) | |
| <b>Interpreter (if required)</b> | 1 | |
| Name of interpreter (if p | oresent): | |
| ID number (if phone into | erpreter): | |
| (The interpreter's name or ID r | number must be documented in the EMR.) | |

The participant/Legally Authorized Representative must be provided with a signed copy of this form.



LAR relationship to

IRB Number: 20-553 A(7) Approval date: 18-Mar-2024

## **Study Calendar:**

This calendar shows the exams, tests, and procedures that will be done as part of this research study, as well as the tests and procedures that are part of your usual care.

| Exams/tests/procedures | Screening | Treatment | After treatment | | | Follow-up |
|---|---|---|---|---|---|---|
| · | | Up to 4 | Week 2 | Week 6 | Week 12 | Starting 26 |
| | | weeks | | | | weeks after |
| | | | | | | RT, then |
| | | | | | | every 6 |
| | | | | | | months for |
| | | | | | | up to 3 years |
| Medical history, physical | X | | X | X | X | |
| exam, vitals | | | | | | |
| Quality-of-life | X | | X | X | X | |
| questionnaires | | | | | | |
| RCM/OCT imaging | | X (Day 0) | | X | | |
| Radiation therapy | | X | | | | |
| Skin biopsy | | | | X | | |
| Check on your health | | | | | | |
| (medical records review, | | | | | | x |
| phone call, email, or | | | | | | ^ |
| letter) | | | | | | |

